CLINICAL TRIAL: NCT07169344
Title: PROSARC-1. Hypofractionated, 3-week, Preoperative Proton or X-ray Radiotherapy for Patients With Localized Soft Tissue Sarcoma. A Single-arm, Multicenter, Phase II Clinical Trial.
Brief Title: Hypofractionated, 3-week, Preoperative Proton or X-ray Radiotherapy for Patients With Localized Soft Tissue Sarcoma
Acronym: PROSARC-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital of Northern Norway, Tromsø, Norway (Unknown); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Ivar Hompland, Senior Consultant, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 915811
Record Dates: First submitted 2025-08-04; First posted 2025-09-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma (Excluding GIST); Soft Tissue Sarcoma Adult; Soft Tissue Sarcoma of the Trunk and Extremities; Synovial Sarcomas; Leiomyosarcoma; Undifferentiated Pleomorphic Sarcoma (UPS); Myxofibrosarcoma (MFS); Liposarcoma; Pleomorphic Rhabdomyosarcoma
Keywords: Soft tissue sarcoma; proton radiotherapy; x-ray radiotherapy; surgical complications
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Dermatofibrosarcoma; Liposarcoma | interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soft tissue sarcoma (Experimental): All patients will receive either proton radiotherapy or x-ray radiotherapy preoperatively, 2.85 Gy x 15.
  Interventions: Radiation: preoperative; Other: Quality of life; Other: Functional outcome

INTERVENTIONS:
Radiation: preoperative — The radiotherapy will be delivered 2.85 Gy x 15 for both x-ray or proton radiotherapy. A comparative doseplan will decide if the patient will receive proton og x-ray radiotherapy.
Other: Quality of life — Questionnaire
Other: Functional outcome — Questionnaire

SUMMARY:
The purpose of the study is to investigate whether a personalized selection of patients with localized soft tissue sarcoma for preoperative proton radiation therapy can reduce long-term radiation side effects without increasing surgical complications or reducing the effectiveness of the treatment. Two radiation plans will be created for each patient-one for protons and one for photons-and through a national meeting, we will determine which type of radiation therapy each patient will receive. The radiation dose will be the same for both photons and protons.

The primary endpoint is surgical complications 120 days after surgery. Secondary endpoints include overall survival, local recurrence-free survival, disease-free survival, side effects, and quality of life. Furthermore, the study will investigate biomarkers that may predict response to radiation therapy, including changes in the tumor's genetic material (DNA), measurement of various molecules in the bloodstream, and the tumor's appearance on MRI scans.

The study will be conducted in Norway, with a planned inclusion of 110 patients.

DETAILED DESCRIPTION:
The objective of the PROSARC-1 trial is to investigate whether a national personalized approach with proton beam therapy (PBT) to selected soft tissue sarcoma (STS) patients can reduce long-term toxicity without increasing surgical complications or compromising local control. PROSARC-1 is a single arm, open-label, multicenter phase II trial initiated at Department of Oncology, Oslo University Hospital (OUS). The main inclusion criterion is patients with newly diagnosed STS of the head, neck, extremity or trunk wall. The primary endpoint is major wound complications (MVC) occurring within the first 120 days after surgery. We expect to include 110 patients over three years and all patients will be followed for up to five years. All the sarcoma centers in Norway participate in the study: OUS; Haukeland University hospital (HUH); St Olavs Hospital (SOH) and the University Hospital of North-Norway (UNN). The indication for preoperative radiotherapy (RT) will be decided in the sarcoma multidisciplinary (MDT) meeting at each center. For included patients, one X-ray radiotherapy (XRT) and one PBT plan will be made for comparison. A weekly national sarcoma radiotherapy meeting will compare the plans and recommend XRT or PBT treatment based on a careful clinical evaluation, also considering thresholds based on the toxicity grade. The prescribed dose is standard 42.75 Gy in 15 fractions over 3 weeks for both XRT and PBT.

The PROSARC-1 trial includes translational radiomic research, where we aim to elucidate underlying mechanisms related to radiotherapy effect. To facilitate future biomarker studies for personalized therapy we will collect excess tumor tissue, whole blood, plasma and serum.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of informed consent.
2. Histological diagnosis of STS, except rhabdomyosarcoma and Ewing sarcoma. Pleomorphic rhabdomyosarcomas are eligible.
3. Primary tumor localized in head, neck, extremity, girdle and/or trunk wall.
4. Measurable disease according to RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
6. Before patient registration, written informed consent must be given according to national and local regulations.
7. Ability to fill in patient questionnaires and comply with study procedures, including travelling to Bergen or Oslo for PBT.

Exclusion Criteria:

1. Locoregional or distant metastasis as assessed by CT and/or MRI at time of diagnosis. Patients with lung nodules <10 mm of uncertain etiology may be included.
2. Prior or concurrent malignant disease whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of this clinical trial are not eligible. Patients with a history of breast cancer, requiring continued hormonal treatment (e.g. anti-estrogen or an aromatase inhibitor) may be included. Patients with a history of prostate cancer, requiring continued support with luteinizing hormone releasing hormone (LHRH) agonists, with or without androgens, may be included.
3. Previous radiotherapy to the primary tumor region.
4. Patients with pacemakers and/or implanted defibrillators.
5. Administration of systemic cancer therapy (i.e. chemotherapy, targeted therapy or immune therapy) within 14 days prior to the first fraction of radiotherapy.
6. Patients not able to give an informed consent or comply with study regulations as deemed by study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2029-01-26 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Major surgical complications | 120 days from surgery
  The criteria that define a major wound complication include the following:
  * Secondary operation(s) required for wound treatment (e.g. debridement, secondary closure procedures such as rotationplasty, vacuum-assisted closure (VAC), free flaps or skin grafts);
  * Readmission to hospital for wound care;
  * Invasive procedures required for wound care (drainage of hematoma, seroma or infected wound collection);
  * Deep wound packing required at any time (deep packing defined as packing deep to dermis in an area of dehisced wound) to an area of wound measuring at least 2 cm in length;
  * Prolonged dressing changes, including packing of the wound for greater than six weeks from wound breakdown;
  * Repeat surgery for revision of a split thickness skin graft or requirement for wet dressings for longer than four weeks. (It is permissible for a patient to protect a totally epithelialized skin graft with a dry dressing without declaring a major wound complication).

SECONDARY OUTCOMES:
Local recurrence-free survival | Up to five years after radiation therapy.
  Local recurrence-free survival is measured from the date of start of study treatment until date of local relapse as evaluated using RECIST v1.1 or date of death of any cause, whichever occurs first
Disease-free survival | Up to five years after radiation therapy
  is measured from the date of start of study treatment until date of progressive disease as evaluated using RECIST v1.1, date of disease recurrence (local relapse or distant metastasis) or date of death of any cause, whichever occurs first.
Overall survival | Up to five years after radiation therapy
  Overall survival is measured from the date of start of study treatment until date of death of any cause.
Overall response rate, defined as partial or complete response using RECIST v1.1 | Up to five years after radiation therapy
  Radiological response will be assessed using MRI and/or CT of the primary tumor.
Pathological response | Perioperative
  pathological response assessed by: Percentage of residual viable tumor cells; Mitotic index; and percentages of the following components of the resected tumor mass: necrosis, hemorrhage, sclerosis, sclerohyalinosis, fibrohistiocytic reaction with hemosiderin.
Health-related quality of life | Up to five years after radiation therapy
  Change from baseline in EORTC QLQ-C30 scores.
Functional outcome | Up to five years after radiation therapy
  Changes from baseline in Musculoskeletal Tumor Society Rating Scale (MSTS)
Functional outcome | Up to five years after radiation therapy
  Changes from baseline in the Toronto Extremity Salvage Score (TESS).

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Hompland, MD, PhD, Principal Investigator — Oslo University Hospital; Kjetil Boye, MD, PhD, Study Director — Oslo University Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olavs University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided